CLINICAL TRIAL: NCT01610830
Title: Identification of Biomarkers Predictive of Worse Prognosis in Henoch Schonlein Purpura
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: HSPRONOSTIC
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2012-07

CONDITIONS: Purpura, Schoenlein-Henoch
Keywords: Purpura, Schoenlein-Henoch; adults; children; pronostic factors
MeSH Terms: conditions — IgA Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine analysis - Skin and kidney biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: have skin involvement +/- an extra renal disease (arthritis, digestive and/or HSP without renal disease. The absence of renal disease is defined by the absence of hypertension (BP <95th percentile for height in children, BP <140/90 mmHg in adults with no known history of hypertension), the absence of hematuria (<5 RBCs per mm3), the absence of proteinuria (proteinuria <0.1 g/24h) and the absence of renal dysfunction (MDRD> 80 ml / min).
- group B: HSP with renal impairment, defined by the presence of renal dysfunction (calculated clearance <60 ml/min) and/or proteinuria (daily proteinuria greater than 0.3 g) and/or hematuria (more than 5000 RBC per ml or 5 RBC per mm3). We distinguish:
  * Group B1 patients with moderate renal disease if renal biopsy was not indicated or no evidence of histologic severity in renal biopsy (histological classification class 1 or 25)
  * Group B2 patients with severe renal impairment, with signs of histological severity in renal biopsy (class 3, 4 or 5).

SUMMARY:
Henoch Schonlein Purpura (HSP), vasculitis of small vessels with deposits of IgA, is considered by many authors as the systemic form of Berger's disease (IgA-N). IgA-N is characterized by IgA1 deposits in mesangial areas associated with mesangial proliferation. These two diseases remain the leading cause of ESRD by primitive glomerulopathy in Western countries. In recent years, considerable progress has been made in understanding the pathophysiological mechanisms of IgA-N. However, only a high rate of proteinuria at one year or the presence of severe glomerular inflammation on renal biopsy remain predictors of long term renal function. Moreover, the high variability of HSP clinical expression, from few purpura skin lesions that evolve favourably spontaneously, to rapidly progressive renal failure, remains so far unexplained but suggests the existence of individual genetic susceptibility.

In the first part of the study, we will study key factors based on physiopathological data obtained by our laboratory as well as by other groups. The second part of the study concerns genetic factors. Although the candidate genes that may confer a particular susceptibility to the disease, to progress to ESRD or respond to treatment are many, the genes involved in inflammation or controlling renin-angiotensin system are of particular interest.

We will apply these results by studying patients with HSP showing three distinct phenotypes (HSP with isolated cutaneous purpura or associated with minimal or severe renal disease) at diagnosis and after clinical remission.

The purpose of this study is to assess whether the phenotype at diagnosis is associated with the physiological markers and if one of them predicts a pejorative evolution of renal disease at 1 year. Meanwhile, study of polymorphism of selected genes of interest could allow identification of patients with specific genetic susceptibility or with bad prognosis factors who would be thus eligible for specific treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HSP whose diagnosis was confirmed by histology of an active skin lesion, who signed the informed consent form or for minors, signature of the holders of parental authority.

Exclusion Criteria:

* Patients who do not have skin lesions; Patients receiving immunosuppressive drugs or steroids for more than 2 weeks; Patients with another diagnosis (platelets<100,000/mm3, bacterial purpura, other systemic disease);
* Patients unable to understand the protocol, refusing to sign the information form or unable to comply with regular follow-up consultation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children or adults, suffering from biopsy-proven HSP.2 groups:
  1. Skin involvement +/- an extra renal disease (arthritis, digestive and/or other), without renal disease. Absence of renal disease is defined by: absence of hypertension (BP <95th percentile for height in children, BP <140/90 mmHg in adults), absence of hematuria (<5 RBCs /mm3 or < 5000 RBCs/ ml), absence of proteinuria (proteinuria <0.1 g/d) and absence of renal dysfunction (MDRD> 80 ml / min)
  2. Renal impairment, defined by the presence of renal dysfunction (calculated clearance <60 ml/min) and/or proteinuria (daily proteinuria greater than 0.3 g) and/or hematuria.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-01 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Renal prognosis | one time measure after a four hour writing session

CONTACTS AND LOCATIONS:
Overall Officials: Evangeline Pillebout, Md PhD, Principal Investigator — APHP - Hôpital St Louis - Paris 10 - France
Locations (1):
- Nephrology Unit - Hôpital St Louis, Paris, France